CLINICAL TRIAL: NCT06841835
Title: Do the Myths of Sexual Orientation Between Nurses and Nursing Students Affect Their Care Behaviours: a Descriptive Study Aimed At Guiding Policy Development for the Care of Individuals Based on Sexual Orientation
Brief Title: Do Nurse and Student Sexual Orientation Misconceptions Effect Care: This Descriptive Research Intended to Inform Sexual Orientation-based Care Policy
Status: Completed | Type: Observational
Sponsor: Şahide Akbulut (Other)
Responsible Party: Sponsor-Investigator, Şahide Akbulut, BatmanU, Batman University
Organization: Batman University (Other)
Other Study IDs: BatmanU-SBF-ŞA-01
Record Dates: First submitted 2025-02-15; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Nursing; Nursing Students
Keywords: sexual orientation myths; care practices; nursing; nursing students

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Abstract Objective: This study aims to investigate the relationship between sexual orientation myths and caregiving behaviours among nurses and nursing students.

Design: A descriptive cross-sectional study was conducted with a total of 321 students enrolled in nursing departments at two state universities and 120 nurses employed at a state hospital. The participants were interviewed in person to complete the "Descriptive Information Form," "Sexual Orientation Myths Scale," and "Caring Behaviours Scale-24.".

Results: The study determined that sexual orientation myths directly affected care behaviours in both groups and high social perception of sexual orientation myths decreased assurance, knowledge and skills, commitment and respectfulness approaches in patient care. It was determined that the mean scores of SOMS disease perception, etiology, sexual behaviour and social perception sub-scores of nursing students were significantly higher and the CBS-24 knowledge and skill sub-dimension was lower than nurses (p<0.01).

Conclusion: These findings suggest that nurses' and nursing students' myths about sexual orientation have a direct impact on their caring behaviour and highlight the importance of developing health policies and educational programmes that promote safe and confidential care for people of sexual orientation.

DETAILED DESCRIPTION:
The literature contains a limited number of studies investigating the sexual orientation myths held by nurses and nursing students. However, no research has been identified that explores the relationship between myths regarding sexual orientation and nursing care behaviours. This situation prompted the design of the study. This study aimed to determine the relationship between myths regarding sexual orientation and the care behaviours of nurses actively involved in care, education, and counselling services, as well as students preparing for the nursing profession.

Design A descriptive and cross-sectional study was conducted in accordance with the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) guidelines.

Hypotheses Research Questions

* What are the sexual orientation myths and care behaviours of nurses and nursing students?
* Is there a significant difference between the mean scores of both sexual orientation myths and care behaviours of nurses and nursing students?
* Is there a significant difference between the mean scores of sexual orientation myths and care behaviours of nurses and nursing students according to their sociodemographic characteristics?
* Is there a significant relationship between the mean scores of sexual orientation myths and care behaviours of nurses and nursing students?
* Does the mean score of sexual orientation myths of nurses and nursing students predict the mean score of caring behaviours? Sample and Timing This study was conducted between September 1, 2022 and December 31, 2022 with 841 students studying in the nursing departments of the health sciences faculties of two state universities located in the east of Turkey and 654 nurses working in a state hospital. When determining the sample size of the study, it was determined that a minimum of 111 people should be sampled in order to conduct a relationship analysis when calculating the sample size using a type I error of 0.05, 95% power, and d: 0.3 effect size. However, in order to determine the relationship between the variables more clearly, the aim was to reach the entire population, and the study was conducted with a total of 321 students studying nursing and 120 nurses working in a state hospital. The study included nurses and nursing students who agreed to participate and had no missing data.

Instruments The Descriptive Information Form, the Sexual Orientation Myths Scale (SOMS), and the Caring Behaviours Scale-24 were used.

Dependent Variable: Mean scores of the Sexual Orientation Myths Scale (CMYS) and the Care Behavior Scale-24.

Independent Variable: Sociodemographic characteristics of the participants

Procedure All the participating students and nurses were informed about the study and their written informed consent was obtained. The researcher collected the data through face-to-face interviews. It took about 15 minutes to fill in the data collection tools. Additionally, the use of self-reported data collection methods may have introduced bias, potentially skewing the results.

Ethical considerations Ethical approval was obtained from University Research and Publication Ethics Committee (decision date and number: 03 February 2022-32). Institutional permission was obtained from the Dean's Office of the Faculty of Health Sciences of both state universities and the Head Medicine of the state hospital in order to conduct the study. Before starting the data collection process, students and nurses were informed about the purpose of the study, voluntary participation, confidentiality issues, and their right to terminate their participation at any time, and written informed consent was obtained from those who agreed to participate in the study. This study was conducted in accordance with the tenets of the Declaration of Helsinki.

Data Analysis The data analysis was conducted by the Statistical Package for the Social Sciences (SPSS) software program. Descriptive statistics were employed to compute values, percentages, means, and standard deviations. The difference in mean scale scores based on categorical variables was assessed using an independent groups t-test for two groups, a one-way ANOVA, or a Kruskal-Wallis test for more than two groups, dependent on the data's normal distribution. The association between numerical variables was evaluated by Spearman correlation analysis based on the data's normal distribution. Statistical significance p<0.05 was accepted at a 95% confidence interval. The effect size was evaluated according to Cohen's effect size classification. In addition, simple regression analysis was used to evaluate whether the mean SOMS score predicted the mean CBS-24 score.

ELIGIBILITY:
Inclusion Criteria:

* To be an active student in the nursing department of universities
* Working as a nurse in a public hospital
* To agree to participate in the study voluntarily

Exclusion Criteria:

* Those who did not agree to participate voluntarily were excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: To be an active student in the department of nursing at the university and working as a nurse in a public hospital
Sampling Method: Probability Sample
Enrollment: 441 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Sexual Orientation Myths Scale (SOMS) | 3 months
  The scale consists of 19 items organised into five sub-dimensions: illness perception, aetiology, sexual behaviour, social perception, and general appearance. They use a five-point Likert format. The tool consists of a five-point Likert scale. The Likert-type scale has five points, with 1 indicating "never agree" and 5 indicating "strongly agree." The total is obtained by collecting the scores from the scale and sub-dimension components. The scale is without a definitive cut-off point. The scale has no reverse-coded items. A minimum of 19 points and a maximum of 95 points can be achieved on the scale. A higher score on the measure is associated with a higher frequency of myths regarding sexual orientation among individuals. The analysis established the value as 0.874.
Care Behaviours Scale-24 (CBS-24) | 3 months
  The scale includes four sub-dimensions and 24 items and uses a six-point Likert-type structure with scores ranging from 1 (never) to 6 (always). The sub-dimensions consist of assurance (8 things), knowledge and skill (5 items), respectfulness (6 items), and connectedness (5 items). In order to determine the total scale score, the scores of 24 items are collected and divided by 24, resulting in a scale score ranging from 1 to 6. To determine the scores for the sub-dimensions, the item scores within each sub-dimension are collected, and the outcome score is divided by the number of items that produce sub-dimension scores ranging from 1 to 6 points

CONTACTS AND LOCATIONS:
Locations (1):
- Batman University Nursing Department, Faculty of Health Sciences,, Batman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No